CLINICAL TRIAL: NCT05772494
Title: Early Assessment of Activity Limitations, a Basis for Understanding the Need for Sickness Certificate and Rehabilitation. A Randomized Controlled Study of People With Mental Disorders in Specialized Psychiatric Care
Brief Title: Assessment of Activity Limitations, a Basis for Understanding the Need for Sickness Certificate and Rehabilitation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: FK 2022/012285
Record Dates: First submitted 2023-03-01; First posted 2023-03-16 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-03

CONDITIONS: Sick Leave
Keywords: Sick leave; Mental disorders; Occupational Therapy; Activity limitations
MeSH Terms: conditions — Mental Disorders | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: The participants are consecutively assigned to either intervention or control group depending on the time for the next prolonged sick leave period. Participants in the intervention group are invited to an assessment session with an occupational therapist focusing on limitations and enablers in activities related to pre-requisites for returning to work. Participants in the control group receive assessments for sickness certificate according to ordinary routines.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Assessment of activity limitation (Experimental): Assessment and analysis of activity limitation by occupational therapist using 2 registered instruments (SDO and DOA).
  Interventions: Other: Assessment of activity limitations, SDO and DOA
- Control group: treatment as usual (Active Comparator): Assessment of activity limitations according to usual routines
  Interventions: Other: Control group

INTERVENTIONS:
Other: Assessment of activity limitations, SDO and DOA — The assessment is made with two instruments (DOA, SDO), and finally the occupational therapist includes the analysis and summary of activity limitations to the sickness certificate. For comparative reasons the participant will answer to a sociodemographic questionnaire focusing on work situation and sick leave
  Other Names: Satisfaction with Daily Occupations (SDO); A Dialogue About Ability Realted to Work (DOA)
  Arms: Assessment of activity limitation
Other: Control group — All assessments concerning activity limitations are made using usual routines, primarily by the sick-listing physician. For comparative reasons the participant will answer to a sociodemographic questionnaire focusing on work situation and sick leave
  Arms: Control group: treatment as usual

SUMMARY:
In Sweden mental disorders have the highest proportion of sickness absence and sickness spells. One cause for this is proposed as the lack of knowledge on which activity limitations that have an impact on the ability to return to work. Further, there is a knowledge gap concerning the effect of which early measures from the health system, assessments and early rehabilitation interventions, that enables return to work. Such early measures have been proposed to have a more multidimensional perspective, than to solely focus on specific tasks during a work situation.

The aim of the current project is to examine the effect of an early assessment of activity limitations, made by occupational therapists within specialized psychiatric care, at the time for the next prolonged sickness certification. The assessment will be included in the sickness certificate, and results will be compared between the intervention group and a control group. The results are calculated for differences on treatment measures, prevalence of questions from the Social Insurance Agency and changes in the patterns for sick leave spells. Further, the prevalence of activity limitations and the sick listed participants assessments of the effect of the intervention will be presented.

The results are expected to lead to more adequate interventions for the individual regarding support to return to work, better routines for assessment and rehabilitation within the health care system, which in turn can facilitate decisions for sickness benefits and further have an impact on the long sick leave spells concerning mental disorders.

DETAILED DESCRIPTION:
Several individuals diagnosed with mental health disorders get sick-listed, and further, stay within the sick-leave process for a prolonged period. More research has been warranted both concerning how to assess activity limitations and future work capacity when having a psychiatric diagnose, but also when it comes to find suitable measures for supporting individuals to return to work. Such supportive and rehabilitative measures could be situated within the healthcare system, such as specialized psychiatric care. To conduct these measures, both early assessments as well as investigation of the effect of taken measures are needed. The present study concerns an expanded assessment of activity limitations as a basis for possible interventions with a focus on the individuals sick-leave process.

The understanding of work capacity has been proposed as a complex phenomenon, where several perspectives are needed. The contribution from occupational therapist in the teamwork implies being focussed on activity limitations or facilitators in contrast to solely focussing on body functions or symptoms. In the professional vocabular, activities are named occupations, meaning that the actual performance is influenced both by individual experiences and influenced by factors in the environment. Another assumption is that all everyday life occupations are interacting, and thus could have an impact on work capacity.

The purpose with this randomized, controlled trial is to evaluate if an early and expanded assessment made by occupational therapist, and with the use of two validated instruments A Dialogue About Ability Related to Work (DOA) and Satisfaction with Daily Occupations (SDO), can have an impact on choice of interventions, changes in the patterns for sick leave spells as well as prevalence of questions from the Social Insurance Agency (SIA) and the participators evaluation of effects from being part of the project. The chosen instruments are described as complementing each other, where DOA examines an overall summary of prerequisites for work capacity, and SDO adds a broader understanding of a person's occupations in everyday life, including satisfaction and balance between different occupational arenas such as work, un-paid work, leisure etc.

The project will be carried out in specialized, psychiatric teams within the Region Västra Götaland. The aim is to recruit 150 participants (75 to the intervention group and 75 to the control group). The participants will be randomly and consecutively divided into intervention or control group. Inclusion criteria are all patients registered at the chosen psychiatric care centres, in need for their second sickness certificate within the unit. Exclusion criteria are patients with specific diagnosis belonging to another unit within the psychiatric organization, and if the patient is assessed as being in an acute vulnerable situation where the planned intervention could negatively influence the situation. Register follow-ups on health care treatment, sick-leave spells, questions from SIA will be made 6 and 12 months later. The participant questionnaire will be sent 6 months after the intervention. Four studies are planned to evaluate the intervention.

The study is a collaborative project involving Region Västra Götaland. The research team comprise researchers from Göteborg University (C Andersson and K Holmgren) and from Region Västra Götaland (C Melin). The study has been submitted to the Regional Ethical Review Board.

ELIGIBILITY:
Inclusion Criteria:

* All patients registered at the chosen psychiatric care centers, in need for their second or third sickness certificate within the unit.

Exclusion Criteria:

* Patients with specific diagnosis belonging to another unit within the psychiatric organization.
* Patients assessed as being in an acute vulnerable situation where the planned intervention could negatively influence the situation e.g. having suicidal thoughts, or having such language difficulties that an interpreter is needed (which could complicate the understanding of the meaning of the intervention and cause unnecessary worries).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-04-03 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Health care treatments | 6 months after inclusion
  Differences in types of healthcare treatment options between intervention and control group. Comparisons will be made between intervention and control group with regard to registered codes for intervention and codes for professionals responsible for treatment options. Descriptive calculations and comparisons will be made on differences in types of as well as changes in treatment measures within the notified time frame.
Changes in sick leave patterns | 6 months after inclusion
  Differences in number of sick leave periods, full-time or part-time or number of sick leave spells between intervention and control group.
Number of questions from the Social Insurance Agency (SIA) | 6 months after inclusion
  Differences in number of clarifying questions from SIA between intervention and control group.

SECONDARY OUTCOMES:
Participants self-assessed effects of being part of the project | 6 months after inclusion
  Data is gathered by a structured questionnaire covering experiences of treatment, support, and effects on need for sick leave after inclusion. Differences in experiences between intervention and control group will be measured. Questions asked are constructed as multiple choice questions, on an ordinal scale, about being on prolonged sick leave, length of sick leave period, having returned to work or not. Questions are further asked about opinions on the effect of treatment on work ability, support for following steps in vocational rehabilitation and contact with other stakeholders within the work rehabilitation process. These latter questions are answered with a 5-point Likert scale, where 1 is "do not agree" and 5 is "fully agreeing".

CONTACTS AND LOCATIONS:
Overall Officials: Christina Andersson, Principal Investigator — Göteborg University
Locations (1):
- Göteborg University, Institute of Neuroscience and Physiology, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No